CLINICAL TRIAL: NCT02746406
Title: A Human Factor Study To Asses The Usability And Feasibility Of The Peritron+ During Intended Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PLUS-HF-01
Record Dates: First submitted 2016-04-12; First posted 2016-04-21 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-09

CONDITIONS: Urology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peritron+ (Experimental): SMIP assessment using Peritron+, Air-Trap Tubing, and a conventional CIC catheter
  Interventions: Device: Peritron+

INTERVENTIONS:
Device: Peritron+ — Peritron+ device to measure intravesical pressure

SUMMARY:
In a hospital setting, the self-measurement of intravesical pressure (SMIP) assessment will be conducted at full and empty bladder using the Peritron+ and a ruler-based manometry method. In the home setting a human factor/usability study will be conducted to measure the subject's ability to perform a successful SMIP assessment at full and empty bladder with the Peritron+. This study involves the use of the Peritron+, Air-Trap Tubing, a ruler and a clean intermittent catheter (CIC).

ELIGIBILITY:
Inclusion Criteria:

* Children (2 to 18 years old)
* Subjects who perform CIC regularly
* Must be able to understand English instructions (written or oral)

Exclusion Criteria:

* Subjects suffering from symptomatic bladder infection

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peritron+
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Peritron+
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Usability Factors; Simple, Doable, and is Comparable to the Ruler-based Manometry Method Using a Questionnaire and Patient Diary.
Description: Each participant could score between 0 and 39 and the total score range for group is 0 to 195. All questionnaires and patient diary questions were summed across the board for patients to derive a total score for the Arm/Group
Time Frame: Through study completion, an average of 4 days
Measure: Number; unit: participants
Arm/Group | Peritron+
Number analyzed (Participants) | 5
participants | 65

ADVERSE EVENTS:
Arm/Group | Peritron+
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release regarding trial results for a period that is less than 60 days. The sponsor can request changes to the communication.